CLINICAL TRIAL: NCT03216369
Title: Short- and Long-Term Hemodynamic Effects Revealed by Arterial Spin Labeling MRI of Carotid Endarterectomy and Carotid Artery Stenting
Brief Title: Short- and Long-Term Hemodynamic Effects of Carotid Endarterectomy and Carotid Artery Stenting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Chief, Chinese PLA General Hospital
Other Study IDs: CEA/CAS-Radiology-ChinaPLAGH
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Stroke
Keywords: Arterial Spin Labeling; MRI; Perfusion; Carotid artery stenting; Carotid endarterectomy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- carotid artery stenting and carotid endarterectomy: Symptomatic patients with unilateral ICA severe stenosis by magnetic resonance angiography were performed 3D pseudo-Continuous Arterial Spin Labeling MRI before and after CAS and CEA.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI perfusion imaging

SUMMARY:
Carotid artery stenting(CAS) and endarterectomy(CEA) are both important treatment strategy for patients with ICA (internal carotid artery) stenosis. Three dimensional pseudo-continuous arterial spin labeling (pCASL) is a noninvasive perfusion imaging modality to detect reperfusion for recanalization therapy. And it provides information about absolute CBF (ml 100 g-1 tissue min-1) at the brain tissue level. The aim of the present study was to evaluate the series hemodynamic changes in patients who had conducted CAS or CEA by using 3D pseudo-continuous arterial spin labeling (pCASL) to explore the potential pattern of CBF alternation and thus to improve the prevention strategy for hyperperfusion syndrome.

DETAILED DESCRIPTION:
Patients:

Patients with unilateral severe internal carotid artery (ICA) stenosis of stroke eligible were enrolled who underwent CAS vs CEA.All patients underwent previous scan in 7 days before CAS and CEA and consecutive scan once per 24 hours after CAS and CEA.

Baseline characteristics of patients were recorded including age,gender, hypertension, hypercholesterolemia, diabetes melitus, smoking, obesity, qualifying stroke event.

Protocols:

MRI scan protocols T2 weighted image,T1 weighted image,diffusion weighted image(DWI),fluid-attenuated inversion recovery (FLAIR),arterial spin labeling(ASL) with Post labeling delay (PLD) of 2.0s,Territory ASL(TASL)(PLD=2.0s),3-dimensional Fast Spoiled Gradient Echo(3D-FSPGR).

Imaging evaluation：

1. Pseudo-continuous arterial spin labeling (pCASL) with post labeling delay (PLD) of 2.0s evaluation of cerebral blood flow in target downstream territory.
2. FLAIR hyperintensity vascular sign.
3. Collateral pattern assessment by Territorial ASL(TASL) (PLD=2.0s).

Treatment strategy:

Patients were randomly treated by CEA(carotid endarterectomy) or CAS(carotid artery stenting).

Follow up:

Patients were followed up every 24 hours after treatment procedure, and would have a repeat MRI scan after 3 months, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* informed patient's consent for ICA stenting or endarterectomy
* lack of contraindications to MRI
* Symptomatic, unilateral ICA stenosis 70-99%;irrelevant stenosis <50% of contralateral ICA
* TIA or stroke - within 360 days

Exclusion Criteria:

* Intracranial hemorrhage
* Informed consent not obtained
* Common exclusion for MRI such as patients with claustrophobia
* Patients with poor imaging quality（Poor imaging quality mainly defined as the image cannot be applied to future analysis on account of severe motion artifacts appeared in conventional MRI and mistakes in the MRI process by accident factors which cannot to be applied to future analysis）
* Bilateral internal carotid artery occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symtomatic patients with unilateral severe internal carotid artery (ICA) stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ischemic Event | Up to 1 year
  The patients will be monitored whether they recured ischemic event including transient ischemic attack (TIA) or stroke confirmed by neurologist and diffusion-weighted image MRI.

SECONDARY OUTCOMES:
Hyperperfusion Syndrome | 3 months
  The patients will be monitored whether they experienced hyperperfusion syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, M.D.,Ph.D., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China